CLINICAL TRIAL: NCT02616354
Title: Preliminary Research On Two-step Dosing Of Imipenem/Cilastatin
Acronym: PROTDOI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jianfeng Xie, Deputy director of the physician, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Two-step Dosing Of Imipenem
Record Dates: First submitted 2015-11-13; First posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Sepsis
Keywords: Pharmacokinetics; pharmacodynamic; imipenem; sepsis
MeSH Terms: conditions — Sepsis | interventions — Imipenem

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Active Comparator): Group I received intravenous imipenem/cilastatin 1 g every 8 h (q8h) or 0.5g every 6 h (q6h) with optimized two-step infusion therapy (OTIT; rapid first-step infusion in 30 min and slow second-step infusion above 1.5 hours) "Group I" is more informative than "Group II" from PK parameters(%T>MIC,AUC/MIC).
  Interventions: Drug: Imipenem
- Group II (Placebo Comparator): group II received intravenous imipenem/cilastatin 1g q8h or 0.5g q6h with extended infusion therapy (2-hours continuous infusion in a constant speed).
  "Group I" is more informative than "Group II" from PK parameters(%T>MIC,AUC/MIC).
  Interventions: Drug: Imipenem

INTERVENTIONS:
Drug: Imipenem — Patients in group I received a dose of imipenem/cilastatin 1g each every 8 hours or 0.5g every 6 hours optimized two-step infusion therapy (rapid first-step infusion in 30 min and slow second-step infusion above 1.5 hours)
  Other Names: Optimized two-step infusion therapy

SUMMARY:
Explore Imipenem/Cilastatin two-step dosing compared to 2 hours infusion in patients with severe whether can obtain better results of the pharmacokinetic/pharmacodynamic, for clinical rational use of antimicrobial agents, and provide theoretical support for optimizing dosage regimen.

DETAILED DESCRIPTION:
Compared with Imipenem/Cilastatin 2 hours continuous dosing method and two-step dosing method (0.5 hours before enter half dose, after 1.5 hours, the other half of the input dose) of blood drug concentration in the body than the minimal inhibitory concentrations (MIC) pathogens percent of dosing interval duration (100% fT > MIC), blood drug concentration in the body more than 4 times the minimal inhibitory concentrations (MIC) pathogens percent of dosing interval duration (100% fT > 4 MIC), blood drug concentration peak and the ratio of the minimal inhibitory concentrations (MIC) pathogens (Cmax/MIC), blood drug concentration (Tmax) used in the peak time, used to guide clinical patients with severe infection of Imipenem/Cilastatin usage.

ELIGIBILITY:
Inclusion Criteria:

* sepsis or severe sepsis or severe infections in the previous 48 hours
* treatment with imipenem/cilastatin (recommended by hospital microbiologists)
* expected duration of hospital stays in the ICU ≥ 72 h from recruitment
* recruited patients agreed to participate in this trial, and had set up a signed informed consent

Exclusion Criteria:

* with an allergy to carbapenems or with an adverse drug reaction to imipenem
* acute or chronic renal failure assessed by serum creatinine concentrations > 280 μmol/L (or creatinine clearance <20mL/min) or those requiring continuous renal replacement therapy
* drug or alcohol abuse
* Pregnant and lactant women
* patients near to death

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | up to 9 months

SECONDARY OUTCOMES:
Plasma Concentration | up to 9 months
  immediately prior to imipenem/cilastatin administration (time 0 min) and at 30 min, 1h, 2h, 4h, 6h and 8h after administration of the infusion

OTHER OUTCOMES:
PK/PD indices | up to 9 moths
  Time>MIC (∫T>MIC) and 4×MIC (∫T>4×MIC)

CONTACTS AND LOCATIONS:
Locations (1):
- Kang Xu, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Huang Y, Xu K, Zhan Y, Zha X, Liu S, Xie J, Liu L, Li Q, Shao H, Yang Y. Comparable Effect of Two-Step Versus Extended Infusions on the Pharmacokinetics of Imipenem in Patients with Sepsis and Septic Shock. Adv Ther. 2020 May;37(5):2246-2255. doi: 10.1007/s12325-020-01339-5. Epub 2020 Apr 10. PMID 32277344